CLINICAL TRIAL: NCT06662461
Title: Efficacy of Ultrasound Guided Block of Stellate Ganglion Versus Greater Occipital Nerve in Chronic Resistant Migraine Patients and Its Correlation to Calcitonin Gene Related Peptide (CGRP)
Brief Title: Ultrasound Guided Block of Stellate Ganglion Versus Greater Occipital Nerve in Resistant Migraine and Correlation to Calcitonin Gene Related Peptide
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Ahmed Mohamed ElSadek (Unknown); Sherien Mohamed Farag (Unknown); Noha Lotfy Soliman (Unknown); Mohamed Amir Tork (Unknown); Ahmed Mohamed Abdelfattah Sharawy (Unknown)
Responsible Party: Principal Investigator, Mai Fathy Ahmed Fahmy, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MD14/2024
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Migraine
Keywords: occipital nerve block; stellate ganglion block; migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound guided bilateral Greater Occipital nerve Block (Active Comparator)
  Interventions: Procedure: ultrasound guided Greater occipital nerve block
- Ultrasound guided bilateral Stellate Ganglion Block (Active Comparator)
  Interventions: Procedure: Ultrasound guided Stellate ganglion block

INTERVENTIONS:
Procedure: ultrasound guided Greater occipital nerve block — Patients will be positioned in a prone position with their neck slightly flexed.
  The trapezius , semispinalis, obliqus capitis muscles will be revealed on short-axis view.
  A 25- or 21 gauge is used, with puncture point 1-1.5 cm away from the ultrasound probe.
  Under the guidance of the ultrasound, GOB will performed by injection using 40 mg triamcinolone and 1ml of 2% lidocaine.
  Arms: Ultrasound guided bilateral Greater Occipital nerve Block
Procedure: Ultrasound guided Stellate ganglion block — Patients are positioned in a lateral position with their necks slightly hyperextended. Assisted by ultrasound imaging equipment the C7 level is confirmed. The thyroid gland, carotid artery, compressible internal jugular vein, vertebral artery, brachial plexus and the oval-shaped structure of the longus collis muscle are revealed on this short-axis view.
  A 25- or 21 gauge is used and the puncture point is 1-1.5 cm away from the ultrasound probe The tip of the needle reach the surface of the longus collis muscle and the 5 o'clock position of the carotid artery. Under the guidance of the ultrasound, SGB is performed by injection using 40 mg triamcinolone and 1ml of 2% lidocaine.
  Arms: Ultrasound guided bilateral Stellate Ganglion Block

SUMMARY:
To investigate the efficacy of Ultrasound guided Stellate Ganglion block in chronic resistant migraine patients in comparison to Greater Occipital Nerve Block correlating its effect to serum CGRP level.

DETAILED DESCRIPTION:
40 Patients diagnosed with Chronic resistant migraine to 2 anti-migraine drugs for 3 months will be evaluated for inclusion and exclusion. Eligible patients with resistance or intolerability to 2 drugs or more will be classified into two groups by using simple randomization methods through Using a computer-generated random number sequence.

Each group will contain 20 patients one group will undergo ultrasound guided bilateral Greater Occipital nerve Block and the other group will undergo ultrasound guided bilateral Stellate Ganglion Block

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with chronic resistant migraine after using or intolerability to 2 or more of anti-migraine drugs for at least 3 months

Exclusion Criteria:

* Patients with a space-occupying lesion.
* Coagulation disorders.
* Systemic or local infection and drug allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Changes in Headache impact test (HIT-6) | 3 months
  Each of the six questions of the HIT-6 receives a score from 6-13. The final HIT-6 score can range from 36 to 78. A higher score indicates more disability due to headache.
changes in Migraine disability assessment test (MIDAS) | 3 months
  The MIDAS questionnaire is based on five disability questions that focus on lost time in three domains: school work or work for pay; household work or chores; and family, social, and leisure activities. The scoring is:
  0-5: little or no disability 6-10: mild disability 11-20: moderate disability 21+: severe disability
changes in Numeric Rating Scale (NRS) | 3 months
  a score used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
Changes in circulating CGRP level | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided